CLINICAL TRIAL: NCT03668964
Title: A Randomized, Double-blinded, Parallel, Placebo-controlled Pilot Study to Investigate the Effect of Nutrition Ingredients on Microbiota Composition in Healthy Adults
Brief Title: Effect of Nutrition Ingredients on Microbiota Modulation
Acronym: VitaGut
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DSM Nutritional Products, Inc. (Industry)
Collaborators: Atlantia Food Clinical Trials (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2017-12-19-VIT
Record Dates: First submitted 2018-05-02; First posted 2018-09-13 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Healthy Volunteers
Keywords: Intestinal microbiota
MeSH Terms: interventions — Riboflavin; Ascorbic Acid; Vitamin A; Cholecalciferol; Vitamin E; alpha-Tocopherol

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, parallel trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Vitamin B2 (Experimental): Daily dose of 75 mg Vitamin B2
  Interventions: Dietary Supplement: Vitamin B2
- Vitamin C (Experimental): Daily dose of 500 mg Vitamin C
  Interventions: Dietary Supplement: Vitamin C
- Vitamin B2 + C (Experimental): Daily dose of 75 mg Vitamin B2 and 500 mg Vitamin C
  Interventions: Dietary Supplement: Vitamin B2 + C
- Vitamin A (Experimental): Daily dose of 250 µg Vitamin A
  Interventions: Dietary Supplement: Vitamin A
- Vitamin D3 (Experimental): Daily dose of 60 µg Vitamin D3
  Interventions: Dietary Supplement: Vitamin D3
- Vitamin E (Experimental): Daily dose of 100 mg Vitamin E
  Interventions: Dietary Supplement: Vitamin E
- Placebo (Placebo Comparator): Daily dose of 575 mg microcrystalline cellulose
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin B2 — One capsule of 75 mg Vitamin B2 once a day for 4 weeks
  Other Names: Riboflavin
  Arms: Vitamin B2
Dietary Supplement: Vitamin C — One capsule of 500 mg Vitamin C once a day for 4 weeks
  Arms: Vitamin C
Dietary Supplement: Vitamin B2 + C — One capsule of of 75 mg Vitamin B2 plus 500 mg Vitamin C once a day for 4 weeks
  Arms: Vitamin B2 + C
Dietary Supplement: Vitamin A — One capsule of 250 µg Vitamin A once a day for 4 weeks
  Arms: Vitamin A
Dietary Supplement: Vitamin D3 — One capsule of 60 µg Vitamin D3 once a day for 4 weeks
  Other Names: Cholecalciferol
  Arms: Vitamin D3
Dietary Supplement: Vitamin E — One capsule of 100 mg Vitamin E once a day for 4 weeks
  Other Names: alpha-tocopherol
  Arms: Vitamin E
Dietary Supplement: Placebo — One capsule of 575 mg microcrystalline cellulose once a day for 4 weeks
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate in healthy volunteers the time-dependent effect of daily consumption for four weeks of six different nutrition ingredients on relative abundance of microbial taxa in fecal samples. Second, the study looks at the time-dependent effect of six different nutrition ingredients on alpha and beta diversity of microbiota in fecal samples. Moreover, the time-dependent effect of six different nutrition ingredients on gastrointestinal symptoms and quality of life will be measured.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects willing and able to give written informed consent and to understand, to participate and to comply with the clinical study requirements;
2. Be between 20 and 50 years of age;
3. Has a BMI of between 18.5 - 30 Kg/m2;
4. Has a stable body weight (< 5% change) over the past 3-months;
5. Is in general good health, as determined by the investigator;
6. Willing to avoid consuming dietary supplements, prebiotic, probiotic, dietary or fibre rich supplements within 4 weeks prior to baseline visit, until the end of the study;
7. Willing to avoid liver consumption during the intervention
8. Maintain current level of physical activity;
9. Women of child-bearing potential using a non-hormonal contraceptive (e.g. IUD);
10. Willing to consume the investigational product daily for the duration of the study.

Exclusion Criteria:

1. Females are pregnant, lactating or wish to become pregnant during the study.
2. Are hypersensitive to any of the components of the test product;
3. Has taken antibiotics within the previous 3 months;
4. Has a history of drug and/or alcohol abuse at the time of enrolment;
5. Consumes greater than 2 servings/day of alcohol (e.g. >28 g ethanol/day);
6. Is a smoker;
7. Has made any major dietary changes in the past 3 months;
8. Subject is planning a sun or ski holiday over the duration of the study;
9. Planned major changes in life style (i.e. diet, dieting, exercise level, travelling) during the duration of the study;
10. Has an eating disorder;
11. Is vegetarian/vegan diet or has food allergies or other issues with foods that would preclude intake of the study products;
12. Is using fibre supplements or enemas;
13. Has a high fiber diet (i.e. >30 g) based on FFQ;
14. Has an active gastrointestinal disorder or previous gastrointestinal surgery,
15. If taking chronic medications (e.g., anti-hypertensive medications), they must have been taking the product for at least two months prior to screening and agree to maintain the same dosage throughout the study;
16. Has a metabolic, psychiatric, or gastrointestinal disease (i.e., diarrhoea, Crohn's disease, ulcerative colitis, irritable bowel syndrome, diverticulosis, stomach or duodenal ulcers, diabetes, hepatitis, HIV, cancer, etc.), with a history of such diseases;
17. Are severely immunocompromised (HIV positive, transplant patient, on antirejection medications, on a steroid for >30 days, or chemotherapy or radiotherapy within the last year);
18. Experiences alarm features such as weight loss, rectal bleeding, recent change in bowel habit (<3 months) or abdominal pain;
19. Have a malignant disease or any concomitant end-stage organ disease;
20. Individuals who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the trial;
21. Subjects may not be receiving treatment involving experimental drugs. If the subject has been in a recent experimental trial, these must have been completed not less than 60 days prior to this study.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Relative abundance of microbial taxa in fecal samples as assessed by shotgun profiling based on shotgun sequencing | from baseline to 4 weeks
  Changes from baseline in the treatment groups as compared to placebo of relative abundance of microbial taxa (operational taxonomic units)

SECONDARY OUTCOMES:
Alpha diversity of microbiota in fecal samples as assessed by shotgun profiling based on shotgun sequencing | from baseline to 4 weeks
  Changes from baseline in the treatment groups as compared to placebo of alpha diversity assessed with shotgun sequencing (Shannon diversity, Estimated ChaoI index)
Beta diversity of microbiota in fecal samples as assessed by shotgun profiling based on shotgun sequencing | from baseline to 4 weeks
  Changes from baseline in the treatment groups as compared to placebo of beta diversity assessed with shotgun sequencing (bray-curtis distance metrics)
Short-chain fatty acids concentrations in fecal samples | from baseline to 4 weeks
  Changes from baseline in the treatment groups as compared to placebo of short-chain fatty acids using GC-MS (mM)
Ammonia concentrations in fecal samples | from baseline to 4 weeks
  Changes from baseline in the treatment groups as compared to placebo of ammonia concentrations assessed with phenol-hypochlorite method (mg/L)
Cytokines and chemokines in blood | from baseline to 4 weeks
  Changes from baseline in the treatment group as compared to placebo of cytokines and chemokines using immune assays (pg/mL)

OTHER OUTCOMES:
Electronic Gastrointestinal Symptom Rating Scale (GSRS) questionnaire | from baseline to 4 weeks
  Changes from baseline in the treatment groups as compared to placebo of the GSRS. The GSRS has a seven-point graded Likert-type scale where 1 represents absence of troublesome symptoms and 7 represents very troublesome symptoms
Short Form 36 (SF-36) questionnaire | from baseline to 4 weeks
  Changes from baseline in the treatment groups as compared to placebo of the quality of life questionnaire Short Form 36 (SF-36) questionnaire. The Short Form (SF)-36 generates a profile of health-related quality of life outcomes by measuring health across eight different dimensions: physical functioning, role limitation because of physical health, social functioning, vitality, bodily pain, mental health, role limitation because of emotional problems and general health. Responses to each question within a dimension are combined to generate a score from 0 to 100; where 100 indicates "good health".
Volatile organic compound levels in fecal samples | from baseline to 4 weeks
  Changes from baseline in the treatment groups as compared to placebo of volatile organic compounds (intensity)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Dinan, Prof, Principal Investigator — Cork University Hospital
Locations (1):
- Atlantia, Cork, Blackpool Cork, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pham VT, Fehlbaum S, Seifert N, Richard N, Bruins MJ, Sybesma W, Rehman A, Steinert RE. Effects of colon-targeted vitamins on the composition and metabolic activity of the human gut microbiome- a pilot study. Gut Microbes. 2021 Jan-Dec;13(1):1-20. doi: 10.1080/19490976.2021.1875774. PMID 33615992